CLINICAL TRIAL: NCT00604955
Title: A Phase 4 Study to Expand Access Program While Assessing the Safety and Efficacy of Paromomycin IM Injection in an Outpatient Setting for the Treatment of Visceral Leishmaniasis
Brief Title: Expand Access/Assess Safety and Efficacy of Paromomycin IM Injection for the Treatment of Visceral Leishmaniasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VLPM03
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Visceral Leishmaniasis
Keywords: visceral leishmaniasis; kala-azar; Bihar, India
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Paromomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Paromomycin IM Injection (approved product in India)
  Interventions: Drug: Paromomycin sulfate

INTERVENTIONS:
Drug: Paromomycin sulfate — Paromomycin will be administered intramuscularly at 11 mg/kg, once a day, for 21 consecutive days
  Other Names: Paromomycin IM Injection

SUMMARY:
This modular Program will first confirm the safety and efficacy of Paromomycin IM Injection when given to an expanded population in the outpatient setting in experienced VL centers and subsequently evaluate the effectiveness of an expanded access model of providing Paromomycin IM Injection to progressively more resource-constrained clinics in Bihar, India.

DETAILED DESCRIPTION:
Safe, effective, and affordable treatments for visceral leishmaniasis (VL) that are widely available to the poorest population of rural India where the disease is endemic are urgently needed. Resistance to antimonials, which have historically been the first line of treatment for VL in Bihar and adjoining states, is a major problem. Other available treatments are limited by their high cost, toxicity, or contraindications in certain populations. Paromomycin IM Injection was approved for the treatment of VL in August 2006 by the Drug Controller General of India (DCGI).

The study is designed to establish a Phase 4 Access Program in a modular, stepwise fashion (Modules 1 to 3). The study will first confirm the safety and efficacy of Paromomycin IM Injection in an expanded VL population treated as an outpatient in experienced centers (Module 1); and then progressively extend the network of treatment facilities, the number and reach of the trained staff, and the implementation of the requisite logistics systems to rural Bihar (Modules 2 and 3). An expanded network of healthcare workers will be trained and supervised to make a preliminary diagnosis of VL; to make appropriate referrals to confirm the diagnosis of VL; to treat with Paromomycin IM Injection; and to assess patient safety and clinical response on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed, newly diagnosed or relapsed visceral leishmaniasis

Exclusion Criteria:

* HIV infection, tuberculosis
* Significant hematologic, renal or liver dysfunction
* Malaria
* Those unable to be treated as an outpatient.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2000 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
M1: Safety as measured by adverse events, serious adverse events, vital signs, and laboratory parameters. | M1: Approximately 6 months
M2&3: Program effectiveness as measured by specific criteria for healthcare workers, patients, and operational systems. | approximately 2.5 years

SECONDARY OUTCOMES:
M1: Clinical cure as measured by temperature/hx of fever, spleen size decrease by at least 33% from baseline, and clinical assessment of treating physician. | M1: Approximately 6 months
M2 and M3: Clinical cure as measured by temperature/hx of fever, spleen size decrease, and clinical assessment of treating physician. | approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: P K Sinha, MD, Principal Investigator — Rajendra Memorial Research Institute of Medical Sciences; T K Jha, MD, Principal Investigator — Kalazar Research Centre; C P Thakur, MD, Principal Investigator — Kala-azar Research Centre; Shyam Sundar, MD, Principal Investigator — Kala-azar Medical Research Centre; Devendra Nath, MD, Principal Investigator — Shrimati Hazari Maternity and Medical Care; Supriyo Mukherjee, MD, Principal Investigator — Research Centre for Diabetes, Hypertension and Obesity; Amrendra K Aditya, MD, Principal Investigator — Dr. A.K. Aditya Clinic
Locations (7):
- India (7):
  - Rajendra Memorial Research Institute of Medical Sciences, Agam Kuan, Patna, Bihar
  - Shrimati Hazari Maternity and Medical Care, Azad Nagar, Balua Tal, Motihari, Bihar
  - Research Centre for Diabetes, Hypertension and Obesity, Bengali Tola, Samastipur, Bihar
  - Dr. A.K. Aditya Clinic, East of Bhola Talkies, Samastipur, Bihar
  - Kala-zar Research Centre, Patna, Bihar
  - Kala-azar Medical Research Centre, Rambagh Road, Muzaffarpur, Bihar
  - Kalazar Research Centre, Brahmpura, Muzaffarpur, Bihar

REFERENCES:
- [Background] Sundar S, Jha TK, Thakur CP, Sinha PK, Bhattacharya SK. Injectable paromomycin for Visceral leishmaniasis in India. N Engl J Med. 2007 Jun 21;356(25):2571-81. doi: 10.1056/NEJMoa066536. PMID 17582067